CLINICAL TRIAL: NCT03766425
Title: Comparison of Efficacy and Safety of Mitomycin and Aflibercept Used to Support Primary Trabeculectomy - a Prospective, Randomized Trial in Patients With Open-angle Glaucoma Undergoing Surgery.
Brief Title: Comparison of Efficacy and Safety of Mitomycin and Aflibercept Used to Support Primary Trabeculectomy.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Justyna Kaproń-Świś, Medical Doctor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/133/2017
Record Dates: First submitted 2018-11-25; First posted 2018-12-06 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Eye Diseases; Optic Nerve Damage; Glaucoma Surgery
Keywords: aflibercept; glaucoma; mitomycin; trabeculectomy
MeSH Terms: conditions — Eye Diseases; Optic Nerve Injuries; Glaucoma | interventions — aflibercept; Mitomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept (Experimental): Aflibercept applied intraoperatively as a subconjunctival injection at a dose of 0.05 ml (40 mg / ml) and one week after the operation at the same dose, also subconjunctival.
  Interventions: Drug: Aflibercept
- Mitomycin (Active Comparator): Mitomycin applied during a surgery at a concentration of 0.3mg / ml for 3 min. on a soaked sponge.
  Interventions: Drug: Mitomycin

INTERVENTIONS:
Drug: Aflibercept — subconjunctival injection
  Other Names: Eylea, Zaltrap
  Arms: Aflibercept
Drug: Mitomycin — subconjunctival injection
  Other Names: Ametycine, Mit-C, Mitomycin C
  Arms: Mitomycin

SUMMARY:
Comparison of efficacy and safety of Mitomycin and Aflibercept used to support primary trabeculectomy - a prospective, randomized trial in patients with open-angle glaucoma undergoing surgery.

DETAILED DESCRIPTION:
Glaucoma is a neurodegenerative disease characterized by progressive dying of retinal ganglion cells, axonal loss and damage to the optic nerve. This leads to a gradual loss of the visual field, and in the final stage to blindness. High intraocular pressure is considered to be the main risk factor for glaucomatous neuropathy. In the treatment we use pharmacological therapies and surgical treatment. The trabeculectomy has been the golden standard for the treatment of glaucoma for many years. This procedure consisting in the creation of a filtering bleb, which allows drainage of aqueous humor from within the eye to underneath the conjunctiva where it is absorbed. in addition to the surgery, anti-proliferative substances play a significant role in suppressing the physiological healing process. Bleb insufficiency observed in the postoperative period results to a large extent from progressive scarring of the follicle, which is responsible for excessive fibroblast proliferation and subconjunctival fibrosis.

Mitomycin is an antineoplastic antibiotic produced by Streptomyces caespitosus. It is one of the bi- or tri-functional alkylating agents causing cross-linking of DNA and inhibition of DNA synthesis. Its properties cause that mitomycin is now a popular medicine used to support trabeculectomy, with proven effectiveness of inhibiting the unwanted healing process of the fistula, and thus extend its period of its proper functioning.

Aflibercept is an inhibitor of vascular endothelial growth factor (VEGF). Its properties cause inhibition of the pathological process of formation of new vessels and their excessive permeability, as well as reduction of leukocyte infiltration and inflammation.

The aim of the research:

Comparison of the effectiveness of primary trabeculectomy in patients with open angle glaucoma supported with Eylea (Aflibercept) compared to the group of patients treated with mitomycin.

Materials and methods:

The research conducted at the Department of Glaucoma Diagnostics and Microsurgery in Medical University of Lublin will include patients treated with antiproliferative substances and trabeculectomy. Two groups of patients will participate in the study:

Group I - patients qualified for mitomycin trabeculectomy Group II - patients qualified for Eylea assisted trabeculectomy (Aflibercept) Mitomycin will be administered in the first group of patients during an operation at a dose of 0.3mg / ml for 3 minutes on a soaked sponge. Aflibercept will be applied intraoperatively in a dose of of 0.05 ml (40 mg / ml) subconjunctival and one week after surgery in the same dose.

Criteria for inclusion:

1. Open angle glaucoma or capsular glaucoma.
2. Patient's age> 40 years
3. Local treatment ineffective due to:

   1. intraocular pressure more than 21mmHg with maximum pharmacological therapy (using B-blocker + carbonic anhydrase + prostaglandins) or
   2. intolerance to topical treatment or
   3. progression in the visual field examination (assessed on the basis of MD, PSD).
4. Lack of previous ophthalmological surgical interventions.
5. No previous laser gonioplasty.
6. No previous laser trabeculoplasty or laser trabeculoplasty performed for more than a year.

Exclusion criteria:

1. Patient with angle-closure glaucoma or secondary glaucoma (except for glaucoma in the course of pseudoexfoliation syndrome).
2. One-eye patient.
3. A patient with pseudophakia or aphakia.
4. Patient after previous ophthalmic procedures (phacoemulsification with intraocular lens implantation, traditional pars plana vitrectomy, keratoplasty).
5. A patient diagnosed or suspected of having uveitis or intraocular inflammation.
6. Any corneal abnormalities or other conditions that make it impossible to reliably test with an applanation tonometer in the treated eye, including earlier refractive surgery of the eye

The efficacy of surgery in both groups will be assessed at subsequent postoperative controls based on the following diagnostic tests:

* Visual acuity examination;
* Intraocular pressure examination;
* Evaluation of the filtering bleb in the slit lamp;
* A photo of the filtering bleb;
* Optical coherence tomography of the filtration bleb;
* Visual field;
* Study of corneal endothelial cell density.

ELIGIBILITY:
Inclusion Criteria:

1. Primary open-angle glaucoma or capsular glaucoma.
2. Patient's age: over 40 years, no sex preference;
3. Local treatment ineffective due to:

   1. Intraocular pressure above 21mmHg at maximum pharmacological therapy (using β-blocker + carbonic anhydrase inhibitor + prostaglandins) or
   2. Intolerance to topical treatment or
   3. Progression in visual field examination
4. Lack of previous ophthalmological surgical interventions.
5. Lack of previously performed laser gonioplasty.
6. No laser trabeculoplasty or laser trabeculoplasty performed for more than a year.

Exclusion Criteria:

1. Patient with primary closed-angle glaucoma or secondary glaucoma (except for glaucoma in the course of pseudoexfoliation syndrome).
2. One-eye patient.
3. Patient with aphakia.
4. Patient after previous ophthalmic procedures (cataract removal by phacoemulsification with an implant of an intraocular lens, vitrectomy by pars plana, keratoplasty).
5. A patient diagnosed or suspected of having uveitis or intraocular inflammation.
6. Any corneal abnormalities or other conditions that prevent reliable testing with an applanation device in the treated eye, including earlier refractive surgery of the eye.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of aflibercept and mitomycin on the morphology of the bleb; | 1 year
  Rating the bleb in The Indiana Bleb Appearance Grading Scale, describing bleb height, extent, vascularity, and leakage with the Seidel test.
Effectiveness of aflibercept and mitomycin on the function of the bleb; | 1 year
  Measurement of intraocular pressure (Goldmann applanation tonometer) and taking a photo of a bleb.

SECONDARY OUTCOMES:
Impact of tested substances on visual acuity after surgery | 1 year
  Examination of a visual acuity 1 week after operation as well as 1 month, 3 months, 6 months, 12 months
The influence of aflibercept and mitomycin on corneal endothelial cell density after surgery | 1 year
  Examination of the corneal endothelial cell density before the surgery as well as 6 months and 12 months after surgery
Impact of used substances on visual field parameters | 1 year
  Examination of a visual field in SITA (Swedish Interactive Testing Algorithm) FAST strategy before the surgery and 12 months after surgery
Frequencies and type of possible complications. | 1 year
  observing and recording all complications and side effects in both groups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Żarnowski, PhD, Study Director — Medical Uniwersity of Lublin al. Racławickie 1 20-059 Lublin; Justyna Kaproń-Swiś, MD, Principal Investigator — Medical Uniwersity of Lublin al. Racławickie 1 20-059 Lublin
Locations (1):
- Medical University of Lublin, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No